CLINICAL TRIAL: NCT02494323
Title: The Evaluation of Dual Channel vs Single Channel FES for Dropfoot
Brief Title: Evaluation of Dual Channel vs. Single Channel FES for Dropfoot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioness Neuromodulation (Industry)
Collaborators: Loewenstein Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Segmented Electrodes
Record Dates: First submitted 2015-03-23; First posted 2015-07-10 (Estimated); Results first posted 2016-04-01 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2015-02

CONDITIONS: Dropfoot
Keywords: Dual Channel Functional Electrical Stimulation; dropfoot, balanced dorsiflexion
MeSH Terms: conditions — Peroneal Neuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Functional Electrical Stimulation (Experimental): Dual channel stimulation of the peroneal nerve to improve dropfoot
  Interventions: Device: Functional Electrical Stimulation

INTERVENTIONS:
Device: Functional Electrical Stimulation — Single channel and dual channel FES for balanced dorsiflexion for patients with dropfoot
  Other Names: Segmented Electrode, Novus System

SUMMARY:
Seventy (70) subjects put on the Ness L300 System, a FES device for ankle dorsiflexion for patients with foot drop. Stimulation will be given through two different electrodes: the QFE which is a single channel stimulation, and the Segmented Electrode which is a dual channel electrode. The purpose of the dual channel stimulation is to enable a balanced dorsiflexion, with no inversion/eversion inclinations. Ankle elevation will be recorded both in a seated position and during gait. Subject preference will be recorded through BSW Questionnaire and Subjective Survey. Twenty first subjects will be stimulated with four different dual channel configurations. The configuration that shows to have an advantage over the others will continue to be evaluated on fifty additional subjects. Same procedure will be taken place, in addition ambulation tests will be performed.

DETAILED DESCRIPTION:
Twenty subjects will be stimulated with a single channel electrode, the Quick Fit Electrode. The values of stimulation will be recorded, as well as ankle movement (balanced Dorsiflexion, inverted or everted Dorsiflexion). Subjects will fill up a Benefit, Satisfaction, Willingness to continue (BSW) form. Next, subjects will be fitted with a segmented Electrode that enables both single and dual channel. Four configurations of current will be compared during sitting position and during gait. The first configuration (A) is segmented electrode single channel stimulation, the second configuration (B) is two currents running in parallel. The first medial channel stimulates the deep branch of common peroneal nerve (dorsiflexion/inversion) and the second lateral current stimulates the superficial peroneal nerve (eversion). In the third configuration (C), channels run diagonally. The medial channel runs between the upper medial electrode and the lateral lower electrode (dorsiflexion/inversion). The lateral channel runs between the lateral upper electrode and the medial lower electrode (eversion). The forth configuration (D) includes a common lower electrode; when it is connected to the upper medial electrode it functions as a medial channel (dorsiflexion/inversion); when it is connected to the upper lateral electrode, it functions as the lateral channel (dorsiflexion/eversion). The subjects will be asked to answer 3 questions after trying each configuration. 1. Thinking of the current system you use, did this test system provide any difference in the way the stimulation feels compared to your existing system? Yes No/Cannot tell any difference. 2. Thinking of the current system you use, did this test system provide any difference in what you think of as the 'quality' of stimulation you are used to compared to your existing system? Yes No/Cannot tell any difference. 3. Thinking of the current system you use, did this test system provide any difference in your ability to walk compared to your existing system? Yes No/Cannot tell any difference After all three dual channel configurations have been tested, subjects will be asked Question 4: Thinking of the last three test systems you used today, which test system do you believe was best among the three? B, C or D Subjects will be asked to grade their satisfaction with the one dual channel system they believe is best using the Benefit, Satisfaction, Willingness to Continue (BSW) questionnaire.

After completing evaluation of the first twenty subjects, a re-evaluation of ten subjects will take place. The anode/cathode electrodes will be re-positioned so the cathodes will be located at the upper part of the cuff and the anodes will be located at the lower part of the cuff. This re-evaluation is needed, since in the first evaluation there was an inconsistency in the anode/cathode positioning in the right and left FES cuffs. Stimulation will be given while sitting and during 2 minutes walk. Ankle movement and stimulation intensity will be recorded and compared to the input received in the initial evaluation of the ten subjects.

Fifty additional subjects were recruited to evaluate the performence of the common anode configuration (configuration D) and compare it to the QFE. configuration D was chosen because it showed an advantage over the other dual channel configurations. Same procedure will take place in order to compare the performance of the Segmented Electrode (configuration D) and the QFE. In addition, ambulation tests will be performed: 2mwt and 10 meter walk test. Gait velocity achieved when using each electrode will be compared to each other and also compared to gait velocity achieved when walking with no stimulation.

ELIGIBILITY:
Inclusion Criteria:• Experienced user or a new user of Functional Electrical Stimulation devices

* Upper motor neuron lesion.
* Foot drop - toe drag during walking.
* Lower limb spasticity- 0-4 according to the modified Ashworth scale.
* Responsible mental state, able to follow multiple step directions.
* Aged between 18 and 80 years old.
* Available for participating in the study.
* Able to understand and sign the informed consent form.
* Able to walk independently or with an assistance device (e.g. cane, walker etc.) / spot guarding for at least 10 meters.
* Ankle passive range of motion preserved between 10 degrees plantarflexion and 30 degrees dorsiflexion.

Exclusion Criteria:

* • Subjects with a demand-type cardiac pacemaker, defibrillator or any electrical or metallic implant.

  * Cancerous lesion of lower limb, present or suspected.
  * Medical condition that prevents participation or would likely lead to inability to comply with the protocol [e.g.: congestive heart failure, patient receiving chemotherapy, uncontrolled epilepsy, etc.].
  * Skin lesion at the site of the stimulation electrodes.
  * Change in bone-joint structures of the lower limb, such as contractures or deformations; fracture or dislocation, which would be adversely affected by motion from the stimulation.
  * Pregnancy.
  * Diagnosis of major depression or psychotic disorder.
  * Participation in another investigation that may directly or indirectly affect the study results.
  * Unable to tolerate electrical stimulation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-03; Primary Completion 2015-06 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bella Kuchuk, Study Director — R&D Clinician
Locations (1):
- Bioness Neuromodulations, Hod HaSharon, Israel

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between 01May to 03Dec2015. Subjects were recruited through Bet-Loweinstein Head Trauma Rehabilitation Department and through Bioness Ltd Clinic Clinic.
Period: Overall Study
Arm/Group | Functional Electrical Stimulation
Started | 70
Completed | 70
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Twenty subjects were evaluated to determine the most advantageous dual channel configuration. When this was determined, 50 additional subjects were evaluated to allow sufficient data do determine feasibility.
Arm/Group | Functional Electrical Stimulation
Number analyzed (Participants) | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (14.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 48
Region of Enrollment [Number; unit: participants]
  Israel | 70

OUTCOME MEASURES:

1. Primary Outcome: Ankle Movement as Good as or Better With the Segmented Electrode as With the QFE
Description: Subjects were fitted with the L300 Cuff that houses the single channel QFE and then the modified cuff that houses the dual channel segmented electrode. Subjects were stimulated first sitting and then after optimal ankle elevation was achieved, they walked with the stimulation. The clinician documented ankle movement on a 5 point scale: 1-inverted dorsiflexion, 2-slightly inverted dorsiflexion, 3-neutral dorsiflexion,4- slightly everted dorsiflexion, 5- everted dorsiflexion. The clinician documented the number of subjects who achieved each movement with each electrode according to the 5 point scale.
Time Frame: 7 months
Population: All subjects suffer from foot drop due to upper motor neuron lesion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Functional Electrical Stimulation
Number analyzed (Participants) | 70
units on a scale | 3.63 (0.85)

2. Secondary Outcome: Benefit Satisfaction Willingness to Continue (BSW) Questionnaire
Description: Number of subjects who benefited or not benefited from the dual channel electrode was counted, number of patients who were satisfied or not satisfied with the dual channel electrode was counted, number of subjects who were willing to continue or who were unwilling to continue with the dual channel electrode was counted
Time Frame: 7 months
Population: Five subjects were excluded from filling up the BSW questionnaire, since the Segmented Electrode (SE) did not produce motor reaction in the ankle
Measure: Number; unit: participants
Arm/Group | Functional Electrical Stimulation
Number analyzed (Participants) | 65
participants
  had benefit from SE | 50
  were satisfied with the SE | 55
  had no benefit from SE | 15
  were not satisfied with the SE | 10
  were willing to continue with the SE | 47
  were not willing to continue with the SE | 18
Statistical Analysis 1: Comparison: Functional Electrical Stimulation; Test type: Superiority or Other; p < 0.01, t-test, 1 sided — P value is adjusted for the comparison of subjects who benefited, were satisfied and willing to continue using the Segmented Electrodes versus subjects who didn't benefit, wern't satisfied ans were not willing to continue using the Segmented Eletrode

ADVERSE EVENTS:
Time Frame: The day of the spot test
Description: Skin was checked for irritation after spot test
Arm/Group | Functional Electrical Stimulation
Serious Adverse Events (participants affected / at risk) | 0/70
Other Adverse Events (participants affected / at risk) | 0/70

LIMITATIONS AND CAVEATS:
A spot test, no time adjusting to stimulation, no home use, indoor environment only, muscle fatigue is an influential factor that was not checked.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days